CLINICAL TRIAL: NCT04604249
Title: Prevalence of COVID-19 and Risk Factors Associated With Seroconversion in La Rinconada, the Highest City of the World - 5,100 m
Brief Title: Prevalence of COVID-19 in High Altitude : Insights From the Highest City of the World
Acronym: RINCOVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre d'Expertise sur l'Altitude EXALT (Other)
Responsible Party: Sponsor
Other Study IDs: RINCOVID
Record Dates: First submitted 2020-10-25; First posted 2020-10-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Covid19; High Altitude
Keywords: Prevalence; Covid-19; SARS-CoV-2; Hight altitude
MeSH Terms: conditions — COVID-19; Altitude Sickness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 rapid diagnostic test (COVID-PRESTO® IgM/IgG, AAZ, Boulogne-Billancourt, France) — Presence of specific SARS-CoV-2 antibodies (IgM or IgG).

SUMMARY:
Since the beginning of 2020, SARS-CoV-2 outbreak spread over the world, conducting in a pandemic state declared by the world health organization in March 2020. Conflicting data have been yet published regarding to the incidence rate of COVID-19 infection in altitude. Mainly based on analysis from national Peru database, some authors argued that COVID-19 disease, as well as case fatality rate was less frequent in altitude. However, epidemiological data are lacking regarding to the prevalence of COVID-19 in altitude, and more specially in high altitude.

Aim of this cross-sectional study is to assess the prevalence of seroconversion for the SARS-CoV-2 in the population of La Rinconada, a mining town at 5,100 m, the highest city in the world.

ELIGIBILITY:
Inclusion Criteria:

- Age > 18 years.

Exclusion Criteria:

* Age < 18 years.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inhabitants of La Rinconda, coming to a medical consultation connected to a scientific research project (Expedition5300).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Prevalence of seroconversion for SARS-CoV-2. | Through study completion, an average of 1 week

SECONDARY OUTCOMES:
2. Occupational and environmental exposures associated with SARS-CoV-2 seroconversion. | Through study completion, an average of 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- La Rinconada, Puno, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castagnetto JM, Segovia-Juarez J, Gonzales GF. Letter to the Editor: COVID-19 Infections Do Not Change with Increasing Altitudes from 1,000 to 4,700 m. High Alt Med Biol. 2020 Dec;21(4):428-430. doi: 10.1089/ham.2020.0173. Epub 2020 Oct 13. No abstract available. PMID 33054403
- [Result] Seclen SN, Nunez-Robles E, Yovera-Aldana M, Arias-Chumpitaz A. Incidence of COVID-19 infection and prevalence of diabetes, obesity and hypertension according to altitude in Peruvian population. Diabetes Res Clin Pract. 2020 Nov;169:108463. doi: 10.1016/j.diabres.2020.108463. Epub 2020 Sep 22. PMID 32971150
- [Result] Segovia-Juarez J, Castagnetto JM, Gonzales GF. High altitude reduces infection rate of COVID-19 but not case-fatality rate. Respir Physiol Neurobiol. 2020 Oct;281:103494. doi: 10.1016/j.resp.2020.103494. Epub 2020 Jul 15. PMID 32679369
- [Result] Woolcott OO, Bergman RN. Mortality Attributed to COVID-19 in High-Altitude Populations. High Alt Med Biol. 2020 Dec;21(4):409-416. doi: 10.1089/ham.2020.0098. Epub 2020 Aug 17. PMID 32815745
- [Result] Intimayta-Escalante C, Rojas-Bolivar D, Hancco I. Letter to the Editor: Influence of Altitude on the Prevalence and Case Fatality Rate of COVID-19 in Peru. High Alt Med Biol. 2020 Dec;21(4):426-427. doi: 10.1089/ham.2020.0133. Epub 2020 Aug 14. No abstract available. PMID 32803989
- [Result] Arias-Reyes C, Zubieta-DeUrioste N, Poma-Machicao L, Aliaga-Raduan F, Carvajal-Rodriguez F, Dutschmann M, Schneider-Gasser EM, Zubieta-Calleja G, Soliz J. Does the pathogenesis of SARS-CoV-2 virus decrease at high-altitude? Respir Physiol Neurobiol. 2020 Jun;277:103443. doi: 10.1016/j.resp.2020.103443. Epub 2020 Apr 22. PMID 32333993
- [Derived] Champigneulle B, Hancco I, Renan R, Doutreleau S, Stauffer E, Pichon A, Brugniaux JV, Pere H, Bouzat P, Veyer D, Verges S. High-Altitude Environment and COVID-19: SARS-CoV-2 Seropositivity in the Highest City in the World. High Alt Med Biol. 2024 Sep;25(3):218-222. doi: 10.1089/ham.2021.0020. Epub 2021 Jul 1. PMID 34197184